CLINICAL TRIAL: NCT05416671
Title: The Effect of Guided Narrative Technique on Child Post-traumatic Stress Symptoms Related to Teachers' Improper Criticism: A Cluster Randomized Controlled Trial
Brief Title: The Effect of Guided Narrative Technique on Child Post-traumatic Stress Symptoms Related to Teachers' Improper Criticism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, YinyinZang, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GNT for Child PTSS
Record Dates: First submitted 2022-05-30; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Posttraumatic Stress Symptoms
Keywords: Children; Teachers' Improper Criticism; Posttraumatic Stress Symptoms; Expressive Writing; Psychological Intervention; Guided Narrative Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Behavioral: guided narrative technique-writing
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: guided narrative technique-writing — The experimental group underwent the psychological intervention of guided narrative technique-writing with the theme of teacher criticism for 20 to 30 minutes once a day for three consecutive days.
  Arms: Treatment group

SUMMARY:
Teachers' improper criticism may lead to posttraumatic stress symptoms (PTSS) in children. This cluster randomized controlled trial examined the effect of guided narrative technique (GNT) on child PTSS caused by teachers' improper criticism in school settings.

ELIGIBILITY:
Inclusion Criteria:

* 5th grade students
* 7-13 years old
* with the ability to read and write

Exclusion Criteria:

* younger than 7 years old or older than 13 years old
* having psychotic disorders

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
change from baseline child posttraumatic stress symptoms at posttreatment | 1 week
  Foa et al.,(2018) revised the Self-Rating Scale for Symptoms of Post-traumatic Stress Disorder in Children (CPSS-5-SR), with Cronbach's α reliability coefficient of 0.78.
  Cpss-5-SR is a 27-item self-reporting measure. Symptom items were scored on a 5-point scale, ranging from 0 (not at all) to 4 (almost always).
change from baseline child posttraumatic stress symptoms at follow-up | 6 months
  Foa et al.,(2018) revised the Self-Rating Scale for Symptoms of Post-traumatic Stress Disorder in Children (CPSS-5-SR), with Cronbach's α reliability coefficient of 0.78.
  Cpss-5-SR is a 27-item self-reporting measure. Symptom items were scored on a 5-point scale, ranging from 0 (not at all) to 4 (almost always).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided